CLINICAL TRIAL: NCT03332264
Title: Sequent Please Drug Coated Balloons Versus Primary Stent Application in Long SFA Lesions
Acronym: SPORTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnoRa GmbH (Industry)
Collaborators: Boston Scientific Corporation (Industry); B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP01
Record Dates: First submitted 2017-10-27; First posted 2017-11-06 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Stenosis; Occlusion; Restenosis
Keywords: PAOD; drug coated balloon; drug coated stent; percutaneous transluminal angioplasty (PTA)
MeSH Terms: conditions — Constriction, Pathologic; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Vessel patency will be compared by quantitative angiography at 12 months in patients who have been treated either with paclitaxel coated balloon catheter, paclitaxel coated stent or bare metal stent in femoropopliteal arteries
Masking Description: Corelab will be masked for the bare metal and paclitaxel coated stent arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug coated balloon catheter (Experimental): PTA with paclitaxel coated "SeQuent Please OTW"
  Interventions: Device: SeQuent Please OTW
- Drug coated stent (Active Comparator): PTA with paclitaxel coated "Eluvia Vascular Stent System"
  Interventions: Device: Eluvia Vascular Stent System
- Uncoated stent (Active Comparator): PTA with bare nitinol stent (as commonly used in site)
  Interventions: Device: Nitinol stent

INTERVENTIONS:
Device: SeQuent Please OTW — Dilatation of occluded or highly stenosed vessel with paclitaxel-coated balloon catheter
  Arms: Drug coated balloon catheter
Device: Eluvia Vascular Stent System — Dilatation of occluded or highly stenosed vessel with paclitaxel-coated stent
  Arms: Drug coated stent
Device: Nitinol stent — Dilatation of occluded or highly stenosed vessel with uncoated bare nitinol stent
  Arms: Uncoated stent

SUMMARY:
Patients with peripheral artery disease will be treated with either drug coated balloon catheter, drug coated stent or uncoated stent.

DETAILED DESCRIPTION:
Patients with chronic stenotic or occlusive atherosclerotic disease and lesions of at least 13 cm length in the SFA or Arteria poplitea segment 1 will be randomized to either treatment with paclitaxel coated balloon catheter, paclitaxel coated stent or bare nitinol stent. Vessel patency will be evaluated by quantitative angiography after 12 months. Clinical follow-ups will be done until 36 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* PAOD and Rutherford classes 2 - 4 (pain-free walking distance <500 m)
* eligible for peripheral revascularization by means of PTA
* peripheral lesions in the superficial femoral artery (SFA) and / or the PI-segment of the popliteal artery (A.pop.)
* minimum diameter stenosis of ≥70%
* treatment length at least 15 cm (lesion length at least 13 cm)
* maximum of lesions to be treated should be 2 (all treated lesions should be treated within the randomization to the study group, i.e. either coated balloon catheters or coated stents or bare nitinol stents); in case of two lesions matching the eligibility criteria, the one presenting the worst attributes (length and stenosis degree) should be chosen as target lesion
* long diffuse stenosis with or without occlusions may only be divided in separate lesions if non-stenotic (i.e. <50% stenosis) segments in between the lesions extent to >2 cm, otherwise vessel segments will be treated as a single extended lesion
* eligible for an operative vascular intervention in case of complications during the PTA

Exclusion Criteria:

* Rutherford class 1,5 or 6
* more than two stenotic lesions in the target vessel requiring treatment
* inflow lesion (proximal to the study lesion) with flow limitation not being successfully treated prior to the study lesion
* in-stent restenosis of the study lesion
* strongly calcified lesions with circumferential presence of calcifications and a lesion calcification length of >4 cm
* reference vessel diameter <4 mm and >6 mm
* guide wire could not be successfully advanced across the lesion
* lesions below the knee requiring treatment
* target lesion is located in the PII-segment of the popliteal artery (A.pop.) or within a bypass graft
* acute thrombosis of the study lesion requiring lysis or thrombectomy prior to the treatment of the study lesion
* potential loss of leg due to critical or acute ischemia
* no patent distal run-off vessel
* medical reason against double anti-platelet therapy in anti-coagulated patient, e.g., receiving coumarine or conditions which prevent the intake of the double anti-platelet therapy for two months
* female patient who is pregnant or lactating
* under 18 years of age
* patients under administrative or judicial custody (§20 Act on medical Devices, Germany)
* expected life span of less than 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Percent diameter stenosis at 1 year post intervention in successfully treated patients | 12 +/- 2 months
  by quantitative angiography

SECONDARY OUTCOMES:
Late Lumen Loss | 12 months
  by quantitative angiography
Binary restenosis | 6,12, 24, 36 months
  by DUS
Target lesion revascularization | 6, 12, 24, 36 months
  number of re-interventions at target lesion

OTHER OUTCOMES:
Event-free survival | 6, 12, 24, 36 months
  absence from target lesion revascularization, amputations and death
Walking distance | 6, 12, 24, 36 months
  assessed in m and compared to baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, MD, Principal Investigator — RoMed Klinikum Rosenheim
Locations (10):
- Medizinische Universität Graz, Graz, Austria
- Germany (9):
  - RoMed Klinikum, Rosenheim, Bavaria
  - Klinikum Arnsberg, Karolinen-Hospital, Arnsberg
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Ihre-Radiologen Standort Franziskus-Krankenhaus, Berlin
  - Ihre-Radiologen Standort Jüdisches Krankenhaus, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Diakonissenkrankenhaus Flensburg, Flensburg
  - SANA Kliniken Lübeck, Lübeck
  - Universitätklinikum Lübeck, Lübeck